CLINICAL TRIAL: NCT03025594
Title: Gonyautoxins Local Periarticular Injection for Pain Management After Total Knee Arthroplasty: A Double Blind Randomized Study
Brief Title: Gonyautoxins Local Periarticular Injection for Pain Management After Total Knee Arthroplasty
Acronym: Toxin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: maximiliano barahona vasquez (Other)
Responsible Party: Sponsor-Investigator, maximiliano barahona vasquez, MD, MBiostat, University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIC 769/15
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Knee Arthroplasty; Pain Management
Keywords: Paralytic sellfish toxins; Gonyautoxin; Post surgery pain management; total knee arthroplasty
MeSH Terms: conditions — Agnosia | interventions — gonyautoxins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gonyautoxin (Experimental): Gonyautoxin 40mcg
  Interventions: Drug: Gonyautoxins
- Control (Active Comparator): Mix of chirocaine 0,2%, ketorolac and epinephrine..
  Interventions: Drug: Chirocaine ketorolac epinephrine

INTERVENTIONS:
Drug: Gonyautoxins — Periarticular infiltration of 40mcg of Gonyautoxin diluted in 30cc of Sodium Chloride 0.9%, with pH 6.2 and isosmotic. This solution will be administer targeting posterior capsule, both retinaculum, collateral ligaments, quadriceps and patelar tendon and subcutaneous tissue just before wound closure of total knee arhroplasty
  Arms: Gonyautoxin
Drug: Chirocaine ketorolac epinephrine — Periarticular infiltration of 150ml of Chirocaine 2%, 60mg of ketorolac and 0.75mg of epinephrine. This solution will be administer targeting posterior capsule, both retinaculum, collateral ligaments, quadriceps and patelar tendon and subcutaneous tissue jbefore wound closure of total knee arhroplasty.
  Arms: Control

SUMMARY:
The aim of this study is to demostrate the eficcacy in pain control management after total knee arthroplasty of Gonyautoxin. Local administration during surgery of Gonyautoxin before wound closure can achieved better pain control and lower morphin use during hospital stay compared to local administration of chirocaine, ketorolac and epinephrine

ELIGIBILITY:
Inclusion Criteria:

* Patients who required total knee arthroplasty due to knee osteoarthritis ( Kellgren and Lawrence score of 2 or more), with no response to conservative management.
* Without known allergies to the drugs used in the study
* Anesthetic risk: ASA Score 1,2,3.

Exclusion Criteria:

* Obesity, defined as body Mass index over 35
* Previous Knee surgery
* Mellitus diabetes
* Organic brain damage
* Rheumatic Arthritis
* Coagulation deficit
* Liver disease
* Chronic obstructive pulmonary disease
* Chronic consumption of opiods
* Refusal to participate in the study

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
morphine consume | 60hrs post surgery
  total consumption of morphine at 60 hours after total knee arthroplaty
range of motion 1 | 12hours post surgery
  Range of motion of the knee that underwent arthroplasty after 12 hours of surgery

SECONDARY OUTCOMES:
early morphine consume | 1 day after surgery
  total morphine consumption during first 24 hours after total knee arthroplaty
range of motion 2 | 36 hours after surgery
  Range of motion of the knee that underwent arthroplasty at 36 hours after surgery
range of motion 3 | 60 hours after surgery
  Range of motion of the knee that underwent arthroplasty at 60 hours after surgery
time of up and go test 1 | 1 day after surgery
  Difference in speed when performing the "up and go" test, which consists of getting up from a chair walk 3 meters and return to sit in the same chair. Comparision will be made between time achieved at 24 hours after surgery compared to time achieved before surgery.
time of up and go test 2 | 2 days after surgery
  Difference in speed when performing the "up and go" test, which consists of getting up from a chair walk 3 meters and return to sit in the same chair. Comparision will be made between time achieved at 48 hours after surgery compared to time achieved before surgery.
pain visual analague scale 1 | 12 hours post surgery
  pain visual analague scale (scale 0-10) applied at rest and post physioterapy
pain visual analague scale 2 | 36 hours post surgery
  pain visual analague scale (scale 0-10) applied at rest and post physioterapy
pain visual analague scale 3 | 60 hours post surgery
  pain visual analague scale (scale 0-10) applied at rest and post physioterapy

CONTACTS AND LOCATIONS:
Overall Officials: Hinzpeter R Jaime, MD, Principal Investigator — orthopaedic surgeon
Locations (2):
- Chile (2):
  - Hospital San Jose, Santiago, Santiago Metropolitan
  - hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Yes
First, a formal letter must be send to the Ethical Committee of Hospital Clinico Universidad de Chile. If the committee gives its consent, the principal investigator will send IPD to whom request it.

REFERENCES:
- [Background] Manriquez V, Castro Caperan D, Guzman R, Naser M, Iglesia V, Lagos N. First evidence of neosaxitoxin as a long-acting pain blocker in bladder pain syndrome. Int Urogynecol J. 2015 Jun;26(6):853-8. doi: 10.1007/s00192-014-2608-2. Epub 2015 Jan 9. PMID 25571865
- [Background] Rodriguez-Navarro AJ, Lagos M, Figueroa C, Garcia C, Recabal P, Silva P, Iglesias V, Lagos N. Potentiation of local anesthetic activity of neosaxitoxin with bupivacaine or epinephrine: development of a long-acting pain blocker. Neurotox Res. 2009 Nov;16(4):408-15. doi: 10.1007/s12640-009-9092-3. Epub 2009 Jul 28. PMID 19636660
- [Background] Rodriguez-Navarro AJ, Lagos N, Lagos M, Braghetto I, Csendes A, Hamilton J, Figueroa C, Truan D, Garcia C, Rojas A, Iglesias V, Brunet L, Alvarez F. Neosaxitoxin as a local anesthetic: preliminary observations from a first human trial. Anesthesiology. 2007 Feb;106(2):339-45. doi: 10.1097/00000542-200702000-00023. PMID 17264729
- [Background] Garrido R, Lagos N, Lattes K, Abedrapo M, Bocic G, Cuneo A, Chiong H, Jensen C, Azolas R, Henriquez A, Garcia C. Gonyautoxin: new treatment for healing acute and chronic anal fissures. Dis Colon Rectum. 2005 Feb;48(2):335-40; discussion 340-3. doi: 10.1007/s10350-004-0893-4. PMID 15812585
- [Background] Garrido R, Lagos N, Lattes K, Azolas CG, Bocic G, Cuneo A, Chiong H, Jensen C, Henriquez AI, Fernandez C. The gonyautoxin 2/3 epimers reduces anal tone when injected in the anal sphincter of healthy adults. Biol Res. 2004;37(3):395-403. doi: 10.4067/s0716-97602004000300005. PMID 15515965
- [Background] Garcia C, del Carmen Bravo M, Lagos M, Lagos N. Paralytic shellfish poisoning: post-mortem analysis of tissue and body fluid samples from human victims in the Patagonia fjords. Toxicon. 2004 Feb;43(2):149-58. doi: 10.1016/j.toxicon.2003.11.018. PMID 15019474
- [Result] Hinzpeter J, Barrientos C, Zamorano A, Martinez A, Palet M, Wulf R, Barahona M, Sepulveda JM, Guerra M, Bustamante T, Del Campo M, Tapia E, Lagos N. Gonyautoxins: First evidence in pain management in total knee arthroplasty. Toxicon. 2016 Sep 1;119:180-5. doi: 10.1016/j.toxicon.2016.06.010. Epub 2016 Jun 15. PMID 27317871
- [Result] Fan L, Yu X, Zan P, Liu J, Ji T, Li G. Comparison of Local Infiltration Analgesia With Femoral Nerve Block for Total Knee Arthroplasty: A Prospective, Randomized Clinical Trial. J Arthroplasty. 2016 Jun;31(6):1361-1365. doi: 10.1016/j.arth.2015.12.028. Epub 2015 Dec 20. PMID 26810604
- [Result] Chaumeron A, Audy D, Drolet P, Lavigne M, Vendittoli PA. Periarticular injection in knee arthroplasty improves quadriceps function. Clin Orthop Relat Res. 2013 Jul;471(7):2284-95. doi: 10.1007/s11999-013-2928-4. Epub 2013 Mar 21. PMID 23516031
- [Result] Andersen LO, Kehlet H. Analgesic efficacy of local infiltration analgesia in hip and knee arthroplasty: a systematic review. Br J Anaesth. 2014 Sep;113(3):360-74. doi: 10.1093/bja/aeu155. Epub 2014 Jun 17. PMID 24939863
- [Result] Albrecht E, Guyen O, Jacot-Guillarmod A, Kirkham KR. The analgesic efficacy of local infiltration analgesia vs femoral nerve block after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2016 May;116(5):597-609. doi: 10.1093/bja/aew099. PMID 27106963
- [Result] Toftdahl K, Nikolajsen L, Haraldsted V, Madsen F, Tonnesen EK, Soballe K. Comparison of peri- and intraarticular analgesia with femoral nerve block after total knee arthroplasty: a randomized clinical trial. Acta Orthop. 2007 Apr;78(2):172-9. doi: 10.1080/17453670710013645. PMID 17464603
- [Result] Moghtadaei M, Farahini H, Faiz SH, Mokarami F, Safari S. Pain Management for Total Knee Arthroplasty: Single-Injection Femoral Nerve Block versus Local Infiltration Analgesia. Iran Red Crescent Med J. 2014 Jan;16(1):e13247. doi: 10.5812/ircmj.13247. Epub 2014 Jan 5. PMID 24719708
- [Result] Affas F, Nygards EB, Stiller CO, Wretenberg P, Olofsson C. Pain control after total knee arthroplasty: a randomized trial comparing local infiltration anesthesia and continuous femoral block. Acta Orthop. 2011 Aug;82(4):441-7. doi: 10.3109/17453674.2011.581264. Epub 2011 May 11. PMID 21561303
- [Result] Ng FY, Chiu KY, Yan CH, Ng KF. Continuous femoral nerve block versus patient-controlled analgesia following total knee arthroplasty. J Orthop Surg (Hong Kong). 2012 Apr;20(1):23-6. doi: 10.1177/230949901202000105. PMID 22535806